CLINICAL TRIAL: NCT03560921
Title: The Association of NGAL With the Development of Acute Kidney Injury After Stored Red Blood Cells Transfusion in Critically Ill Patients.
Brief Title: Urinary NGAL Acute Kidney Injury After Stored Red Blood Cells Transfusion in Critically Ill Patients.
Status: Completed | Type: Observational
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Tarek Samy Abdelziz, Senior lecturer, Kasr El Aini Hospital
Other Study IDs: KA-13115
Record Dates: First submitted 2018-06-05; First posted 2018-06-18 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Acute Kidney Injury; Anemia
Keywords: biomarkers
MeSH Terms: conditions — Acute Kidney Injury; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stored blood transfusion: measurement of urinary NGAL
  Interventions: Diagnostic Test: urinary NGAL
- Fresh blood transfusion: measurement of urinary NGAL
  Interventions: Diagnostic Test: urinary NGAL

INTERVENTIONS:
Diagnostic Test: urinary NGAL — measurement urinary NGAL using the ARCHITECT technique

SUMMARY:
The study aims to explore the association of the novel urinary bio marker NGAL with the age of PRBCs(packed red blood cells) transfusion in critically ill patients.

DETAILED DESCRIPTION:
The investigators will measure the urinary NGAL in all patients who received blood transfusion in the intensive care unit during the study period. The age of PRBCs transfusion will be correlated with the incidence of AKI. The rise of NGAL and serum creatinine will be used to diagnose AKI (Acute Kidney Injury).

ELIGIBILITY:
Inclusion Criteria:

* Any patients admitted to the intensive care unit.

Exclusion Criteria:

* patients who have established AKI at the time of recruitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to ICU of any age and sex
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2017-12-05 (Actual); Study Completion 2017-12-05 (Actual)

PRIMARY OUTCOMES:
Incidence of AKI | within 30 days
  Diagnosis of AKI by rise of serum creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Abdelaziz, Principal Investigator — faculty of medicine-Cairo University Hospitals
Locations (1):
- Cairo university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No